CLINICAL TRIAL: NCT03120832
Title: Phase 1, Open Label Trial to Evaluate the Safety and Immunogenicity of PAN-301-1 in Cancer Patients
Brief Title: Phase 1 Trial of PAN-301-1 (SNS-301) in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sensei Biotherapeutics, Inc. (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAN0216
Record Dates: First submitted 2017-02-16; First posted 2017-04-19 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PAN-301-1 (SNS-301) Vaccine (Experimental): PAN-301-1 vaccine is administered intradermally in 3 cohorts of patients in a dose escalation schema every 21 days
  Interventions: Biological: PAN-301-1

INTERVENTIONS:
Biological: PAN-301-1
  Other Names: SNS-301

SUMMARY:
This is a Phase I, open-label, parallel design study of PAN-301-1 (SNS-301), a HAAH directed nanoparticle vaccine, given intradermally in cohorts of patients with biochemically relapsed prostate cancer, using a fixed dose escalation schema every 21 days.

DETAILED DESCRIPTION:
Human aspartyl-asparaginyl-β-hydroxylase (HAAH), also known as aspartate-β-hydroxylase, is an ~86 kDa type 2 transmembrane protein that belongs to the α-ketoglutarate-dependent dioxygenase family. It is a highly conserved enzyme, which catalyzes the hydroxylation of aspartyl and asparaginyl residues in epidermal growth factor-like domains of proteins including Notch and homologs. HAAH was initially identified in a novel screen to identify cell surface proteins up-regulated in liver cancer. It has subsequently been detected in a diverse array of solid and blood cancers, including: liver, bile duct, brain, breast, colon, prostate, ovary, pancreas, and lung cancers as well as leukemia. HAAH is not found in significant quantities in normal tissue or in proliferative disorders.

The investigators have designed a bacteriophage lambda system to display HAAH peptides fused at the C terminus of the head protein gpD of phage lambda. The phage carry 200-300 copies of the gpD protein on their head and thus display many copies of an approximately 25 kDa molecular weight fragment of HAAH on their surface. The drug substance is one of these HAAH bacteriophage lambda constructs: HAAH-1λ (PAN-301-1).

This study evaluates the safety and immunogenicity of the PAN-301-1 vaccine in patients with biochemically-relapsed prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Ethics Committee approved informed consent
2. Men aged 21 to 85 years with a histologic diagnosis of prostate cancer with a biochemical relapse following definitive local therapy (RP or radiation therapy)
3. Patients are not eligible or are unwilling to receive additional definitive therapy following relapse (either RP or radiation therapy)
4. No prior cytotoxic chemotherapy for the current cancer
5. Normal electrocardiogram (ECG) or ECG with no clinically significant findings as determined by the Principal Investigator
6. Presence of biochemically relapsed prostate cancer defined as either: 1) PSA > 2 ng/mL 1 year following initial definitive treatment for prostate cancer: or, 2) PSA doubling time (greater than 0.2 ng/mL) < 12 months; or, 3) PSA velocity > 2 ng/mL/year at any time following radical prostatectomy or radiation therapy.
7. Positive expression of HAAH in either archived tumor tissue (if available) or fresh serum
8. No clinical or radiologic evidence of distant metastatic disease as measured by pelvic MRI or CT scan in addition to bone scan. These studies will need to be performed within 56 (+ 7 days) days prior to the start of the study.
9. No history of immunosuppressive disease
10. No evidence of active autoimmune disease. Active autoimmune disease is defined as any disease process that has specifically needed administration of immune suppressive and or cytoreductive therapy currently or within the last 1 year.
11. Able and willing to comply with all study procedures

Exclusion criteria:

1. PSA doubling time of < 3 months
2. Participation in a clinical trial within 30 days prior to enrollment
3. Prior major surgery or radiation therapy within 4 weeks of enrollment
4. Any illness or condition that in the opinion of the Investigator may affect the safety of the patient or the evaluation of any study endpoint
5. Screening blood counts of the following:

   Hematopoietic:

   Absolute neutrophil count < 1500/μL, Platelets < 100,000/μL, Hemoglobin < 9 g/dL;

   Liver/Metabolic:

   Alanine aminotransferase (ALT) and aspartate transaminase (AST) > 2.5 × ULN range, Total bilirubin > 2 × ULN, Albumin < 2.8 g/dL;

   Renal:

   Creatinine clearance < 50 mL/min as predicted by the Cockcroft-Gault formula
6. Subjects whose partners are WOCBP must use an adequate method of birth control while on study drug and at least for 3 weeks after discontinuation of study drug
7. Current or anticipated concomitant immunosuppressive therapy (excluding nonsystemic inhaled, topical skin and/or eye drop-containing corticosteroids)
8. Any concurrent condition requiring the continued use of systemic steroids (see above) or the use of immunosuppressive agents including methotrexate. All other systemic corticosteroids must be discontinued at least 4 weeks prior to first study treatment
9. Receipt of any blood product within 1 month of enrollment
10. Receipt of any vaccine within 4 weeks of enrollment
11. Active drug or alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirements
12. Been imprisoned or compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infectious disease) illness
13. Patients who have a history of coagulopathies, thrombosis or who are receiving active anticoagulation for any condition, such as but not limited to, artificial heart valves, atrial fibrillation, etc.
14. Any other conditions judged by the Investigator that would limit the evaluation of a subject

Ages: 21 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be male subject having diagnosis of prostate cancer
Enrollment: 12 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Urology Centers of Alabama, Homewood, Alabama
  - Dr. James J. Elist, Beverly Hills, California
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: PAN-301-1 vaccine is administered intradermally in 3 cohorts of patients in a dose escalation schema every 21 days In this cohort it is administered as SNS-301 2.0 x 10^10 particles/administration intradermally once every 21 days. Then from 6th treatment visit escalated within same patient to dose 10^11 particles/administration intradermally once every 21 days. Then from 11th treatment visit escalated within same patient to dose 3 X 10^11 particles/administration intradermally once every 21 days.
- Cohort 2: PAN-301-1 vaccine is administered intradermally in 3 cohorts of patients in a dose escalation schema every 21 days In this cohort it is administered as SNS-301 1.0 x 10^11 particles/administration intradermally once every 21 days. Then from 6th treatment visit escalated within same patient to dose 3 X 10^11 particles/administration intradermally once every 21 days.
- Cohort 3: PAN-301-1 vaccine is administered intradermally in 3 cohorts of patients in a dose escalation schema every 21 days In this cohort it is administered as SNS-301 3.0 x 10^11 particles/administration intradermally once every 21 days.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 3 | 2 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (1.73) | 67 (6.24) | 72.8 (9.62) | 69.9 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 1 | 3 | 6 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed by Development of Adverse Events and Dose-limiting Toxicity to Determine Maximum Tolerated Dose
Time Frame: Through the 21 day interval after the first dose of vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 6
Participants
  No Dose Limiting Toxicity Observed | 3 | 3 | 6
  Dose Limiting Toxicity Observed | 0 | 0 | 0
  Maximum Tolerated Dose Reached | 0 | 0 | 0

2. Secondary Outcome: Safety Assessed by Administration Site Reactions, Abnormal Laboratory Values and/or Adverse Events
Time Frame: Through study completion, an average of 3 months. Patients were able to continue on treatment with one patient receiving approximately 15 months of treatment.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 6
Participants
  Subjects with no treatment related adverse events observed | 2 | 1 | 6
  Subjects with treatment related adverse events observed | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 months after last dose/visit, a total of about 640 days since the start of the study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypochloremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis hemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT03120832/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03120832/SAP_001.pdf